CLINICAL TRIAL: NCT04893850
Title: Building Regulations in Dual Generations at KIDTHINK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Leslie E. Roos, Assistant Professor Departments of Psychology and Pediatrics, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRIDGE KIDTHINK
Record Dates: First submitted 2021-05-14; First posted 2021-05-20 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2021-06

CONDITIONS: Depression; Child Development; Self-regulation
MeSH Terms: conditions — Depression; Self-Control

STUDY DESIGN:
Intervention Model Description: The study will recruit a group of caregivers in which the caregiver meets the current criteria for elevated symptoms of psychological distress as measured by a score of 9 and above on the Patient Health Questionnaire 9-item. Eligible caregivers (mothers, fathers, guardians) will be randomly assigned to one of two intervention arms, which will occur concurrently over 16-weeks. One arm will incorporate intervention materials from Dialectical Behavior Therapy (DBT) and parent skills training, while another will provide community family support services as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BRIDGE-KIDTHINK Condition (Experimental): Caregivers in this group will participate in 16 sessions of online therapy delivered through a combination of asynchronous material and virtual support groups. These sessions will include Dialectical Behaviour Therapy (DBT) and parenting training. This group will be asked to evaluate the program with surveys completed pre-program, immediately post-program, and three months post-program. This group will also be invited to complete weekly surveys expected to take 5 minutes.
  Interventions: Behavioral: BRIDGE Therapy Program
- Services as Usual Condition (Experimental): Caregivers in this group will not participate in Dialectical Behaviour Therapy (DBT) and parenting training. Rather, this group will be asked to refer to a list of community mental health and family support services as part of the BRIDGE therapy program. This group will be asked to complete weekly surveys expected to take 5 minutes.
  Interventions: Behavioral: Community Services as Usual Clinical Referral list

INTERVENTIONS:
Behavioral: BRIDGE Therapy Program — The BRIDGE Therapy Program is a novel manualized therapy that incorporates key parenting concepts and related Dialectical Behavior Therapy (DBT) modules. The primary aim of the program is to improve parent well-being and promote supportive parenting practices. There are two components of the program: 1) the DBT section, which will follow the DBT Skills Training Manual 2nd Edition and target parental mental health symptomology, and 2) the parent skill training materials, which have been designed to correspond to the four core DBT modules (i.e., Mindfulness, Emotion Regulation, Distress Tolerance, and Interpersonal Effectiveness) and to promote self-regulatory skill development and a positive parent-child relationship.
  Arms: BRIDGE-KIDTHINK Condition
Behavioral: Community Services as Usual Clinical Referral list — The community services as usual clinical referral list provides information on accessing psychological and family support services in Winnipeg. This resource is used to locate: crisis, distress, and support phone lines, counselling and peer-support resources, and free apps relating to mindfulness and meditation.
  Arms: Services as Usual Condition

SUMMARY:
Neurodevelopmental disorders (NDDs) such as attention deficit hyperactivity disorder (ADHD), autism spectrum disorder (ASD), and intellectual disability (ID) are the most frequently diagnosed disability in children, accounting for 7% to 14% of children in developed countries. Developmental concerns emerge early, providing an opportunity to support families years before a diagnosis may occur. Emerging concerns are often predictive of problems with self-regulation, risky behaviours (e.g., substance abuse and over-eating), academic achievement, social functioning, parent-child relationship, and lower overall quality of life. Overall family wellbeing is also commonly affected given the increased challenges faced by parents and caregivers, including socioeconomic disadvantage. Parents facing hurdles to positive parenting, such as poor psychological wellbeing, may struggle further with parenting capacity in the context of the increased parenting demands of caring for a child with specific needs. The objective of this study is to create a novel adaptation of an existing program that is targeted at improving the mental wellness and parenting practices of caregivers (mothers, fathers, guardians) with elevated symptoms of depression who have 3 to 8-year-old children with emerging behavioural, emotional, or developmental concerns. It is hypothesized that taking a dual-generation intervention approach to addressing self-regulatory mechanisms underlying psychopathology at the level of the caregiver, child, and dyad (i.e. parenting interactions) will improve both caregiver capacities and child outcomes. Further, it is hypothesized that this novel adaptation of the program will be tailored to meet the identified needs of this demographic and that the program will show improvement in psychosocial, emotional, and parenting function compared to a services as usual control group. Our current study will be conducted remotely due to the COVID-19 pandemic to adhere to public health guidelines to reduce in-person contact and physical distance. The ultimate goal of this project is to improve parent wellbeing and promote supportive parenting practices that allow children with early developmental needs to reach their full potential.

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregivers must have a 3-8 year old child.
* The child must have diagnosed or emerging behavioural, emotional, or developmental concerns, as reported by parents.
* Parents/caregivers must be experiencing elevated symptoms of psychological distress as measured by the Patient Health Questionnaire 9-item (PhQ-9).
* Parents/caregivers must be 18 years of age.

Exclusion Criteria:

* Child is outside of the 3-8 year old age range.
* The child does not have diagnosed or emerging behavioural, emotional, or developmental concerns.
* The parent or caregiver does not have full or joint custody of the child.
* The parent or caregiver is not experiencing elevated symptoms of psychological distress as measured by the Patient Health Questionnaire 9-item (PhQ-9).
* The parent or caregiver is not 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
Changes in the Child Behaviour Checklist (CBCL) from pre-intervention to post-intervention. | The Child Behaviour Checklist will be completed by participants at baseline prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 16 weeks after baseline).
  99-item questionnaire used to measure child functioning across internalizing/externalizing problems. Participants respond to items on a 3-point Likert scale and are asked to describe their child's behavioural and emotional problems within the past 2 months.
Changes in the Life Events Checklist (LEC) from pre-intervention to post-intervention. | The Life Events Checklist will be completed by participants at baseline prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 16 weeks after baseline).
  34-item measure that assesses adverse life experiences of children.
Changes in Child Functioning from pre-intervention to post-intervention. | Open-ended questions regarding child functioning will be completed by participants at baseline prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 16 weeks after baseline).
  Open-ended questions regarding child functioning for qualitative analysis.

SECONDARY OUTCOMES:
Changes in parent/caregiver emotion regulation from pre-intervention to post-intervention - Difficulties in Emotion Regulation Scale (DERS-16). | The Difficulties in Emotion Regulation Scale will be completed by participants at baseline prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 16 weeks after baseline).
  16-item measure that assesses emotional regulation, including awareness, clarity, goals, impulsivity, nonacceptance, and regulation strategies. Participants respond to items on a 5-point Likert scale. Higher scores suggest more severe problems with emotion regulation. The highest possible score is 80 and the lowest possible score is 16.
Changes in parenting/caregiving stress from pre-intervention to post-intervention - Parenting Stress Index (PSI; Short form). | The Parenting Stress Index will be completed by participants at baseline prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 16 weeks after baseline).
  36-item self-report measure filled out by parents to measure stress level within the context of parenting. Participants respond to items on a 5-point Likert scale. There are 3 sub categories. Responses to each item in a sub-category are totalled and then the 3 subcategory scores are summed to represent a total stress score. Higher scores indicated higher levels of parenting stress. Normal scores fall within the 15th to 85th percentile, and scores above the 85th percentile represent clinically elevated levels of stress.
Changes in recent stressful events from pre-intervention to post-intervention - Recent Stressful Events (RSE). | The Recent Stressful Events Measure will be completed by participants at baseline prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 16 weeks after baseline).
  Assesses the frequency of stressful events in the past month and past year. Developed based on recommendations from the JBP research network on toxic stress at the Harvard's Center on the Developing Child.
Changes in parental/caregiver depressive symptoms throughout the intervention - Patient Health Questionnaire - 9 (PHQ-9). | The Patient Health Questionnaire - 9 will be completed by participants weekly throughout the intervention (approx. 16 times throughout 16 weeks).
  A measure that assesses depressive symptoms using 8-items that align with diagnostic criteria. For the purposes of this study item 9 (regarding suicide ideation) will not be used.
Changes in parental/caregiver perception of social support from pre-intervention to post-intervention - Multidimensional Scale of Perceived Social Support (MSPSS). | The Multidimensional Scale of Perceived Social Support will be completed by participants at baseline prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 16 weeks after baseline).
  A 12-item measure that assesses perceived social supports in parents/caregivers. Participants respond to items on a 7-point Likert scale. Higher scores are indicative of increased perception of social support.
Changes in parenting/caregiving quality from pre-intervention to post-intervention - Coping with Children's Negative Emotions Scale (CCNES). | The Coping with Children's Negative Emotions Scale will be completed by participants at baseline prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 16 weeks after baseline).
  A measure with 12 items (each with 6 sub-items for a total of 72 responses) that assesses parenting quality across supportive and unsupportive dimensions. Participants respond to items on a 7-point Likert scale.
Changes in perceived parental/caregiver resilience from pre-intervention to post-intervention - Connor-Davidson Resilience Scale 2 (CD-RISC 2). | The Connor-Davidson Resilience Scale 2 will be completed by participants at baseline prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 16 weeks after baseline).
  A 2-item measure that assesses self-reported resilience over the past month. Participants respond to items on a 5-point Likert scale. Higher scores are indicative of increased perceived resilience.
Changes in various aspects of parenting/caregiving from pre-intervention to post-intervention - Parenting Scale (PS). | The Parenting Scale will be completed by participants at baseline prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 16 weeks after baseline).
  A 30-item measure that assesses various aspects of parenting, including overreactivity, laxness, and verbosity. Participants are asked about their parenting style during the past two months.
Changes in parental/caregiving spanking from pre-intervention to post-intervention - Parental Spanking. | The Parental Spanking Measure will be completed by participants at baseline prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 16 weeks after baseline).
  A single-item measure assessing the frequency of spanking on a child's bottom during a typical year (restricted to age 2-5 years due to mandatory reporting guidelines for child maltreatment).
Changes in family resources from pre-intervention to post-intervention - Family Resource Scale - Revised (FRS-R). | The Revised Family Resource Scale will be completed by participants at baseline prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 16 weeks after baseline).
  A 29-item measure assessing whether families have adequate resources to meet the needs of the family as a whole as well as individual needs within the family. Participants respond to items on a 6-point Likert scale.
Changes in marital functioning from pre-intervention to post-intervention - Revised Dyadic Adjustment Scale (RDAS). | The Revised Dyadic Adjustment Scale will be completed by participants at baseline prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 16 weeks after baseline).
  A 14-item measure that assesses marital functioning across three subscales: cohesion, consensus, and satisfaction. Participants respond to items on a 6-point Likert scale.
Changes in Parental/Caregiver Functioning from pre-intervention to post-intervention. | open-ended questions regarding parent/caregiver functioning will be completed by participants at baseline prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 16 weeks after baseline).
  Open-ended questions regarding parental/caregiver functioning and unmet needs.

OTHER OUTCOMES:
Changes in child socioemotional and behavioural functioning from pre-intervention to post-intervention - Strengths and Difficulties Questionnaire (SDQ). | The Strengths and Difficulties Questionnaire will be completed by participants at baseline prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 16 weeks after baseline).
  A 25-item measure that assesses child and socioemotional behavioural functioning over the last six months or current school year. Parents/caregivers respond to items on a 3-point Likert scale.
Changes in specific parenting/caregiving behaviours and strategies - Parenting Young Children (PARYC). | The Parenting Young Children Measure will be completed by participants at baseline prior to the beginning of the BRIDGE Therapy Program and at Time 2 once again after the program is complete (approx. 16 weeks after baseline).
  A 21-item measure assessing specific parenting behaviours and strategies during the last month. Parents/caregivers respond to items on a 5-point Likert scale.
Changes in parent/caregiver reports of child behaviours - Parent Daily Report - Revised Version. | The Revised Parent Daily Report will be completed by participants weekly throughout the intervention (approx. 16 times throughout 16 weeks).
  Parent/caregiver reports of child behaviours in the past 24 hours. Participants respond to items on a 3-point Likert scale indicating whether a thought/behaviour occurred for their child, and whether it was stressful for them as the parent/caregiver.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Manitoba - Department of Psychology, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No